CLINICAL TRIAL: NCT00704587
Title: Flow Cytometrical Analysis of the Human Immune System to Assess Tumor-related Material Piling up in Activated Macrophages in All Relevant Cancer Types.
Brief Title: Prognostic Factors for All Types of Cancer Combined
Acronym: ProFaCo
Status: Completed | Type: Observational
Sponsor: Atrium Medical Center (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Dennis Japink, drs, Atrium Medical Center
Other Study IDs: ProFaCo; METC 06-p-47; MEC 08-02-030; NL14215.096.06
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Cancer
Keywords: cancer occurence; cancer recurrence; neo-adjuvant treatment response measurement
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — white cells
  tissue
  plasma
  serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate every possible applicability of flow cytometrical analysis in the intracellular detection of tumor-related material in activated macrophages in the broadest range of cancer types.

ELIGIBILITY:
Inclusion Criteria:

* (Suspicion of) presence of cancer in the broadest sense of the word
* Must be able to understand and sign written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients diagnosed or suspected of cancerous conditions in the broadest sense of the word
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2006-11; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
screening and followup | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Japink, MD, Principal Investigator — Atrium Medical Centre Parkstad, Heerlen
Locations (2):
- Netherlands (2):
  - Atrium Medical Centre Parkstad, Heerlen, Limburg
  - Maastricht University Medical Centre, Maastricht, Limburg